CLINICAL TRIAL: NCT05530447
Title: An Intermediate-size, Expanded Access to SUVN-G3031 for the Treatment of Subjects With Narcolepsy Who Have Completed the CTP2S13031H3 Protocol
Brief Title: Expanded Access to SUVN-G3031 (Samelisant) for the Treatment of Subjects With Narcolepsy
Status: No longer available | Type: Expanded Access
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP13031H3
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — samelisant

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Samelisant — Tablet
  Other Names: SUVN-G3031

SUMMARY:
The study is planned to provide expanded access treatment to subjects with narcolepsy who have completed the 2-week treatment phase and follow-up in study CTP2S13031H3 (NCT04072380), and in instances when the investigator as well as the subject believe that the benefits outweigh the risks to continue the treatment with SUVN-G3031.

DETAILED DESCRIPTION:
The qualified subjects will be given 2mg of SUVN-G3031 expanded access treatment for 30 days. At the end of 30 days if the subject wishes to continue the treatment, he/she will be provided with adequate investigational drug for next 30 days. This cycle will be repeated up to a maximum of 2 times (total duration of expanded access treatment up to 90 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed the 2-week treatment phase and follow-up period of study CTP2S13031H3 (NCT04072380) as planned and wish to continue unblinded treatment with SUVN-G3031 (2 mg, qd).
2. Subject must sign the ICF to participate in the study.
3. The investigator after review of relevant information and in consultation with the subject believes that continued treatment following study CTP2S13031H3 could be beneficial to the subject.

Exclusion Criteria:

1. Any clinically relevant concomitant disease or AEs/SAEs during the Phase 2 study (CTP2S13031H3), which in the opinion of the investigator, makes the subject unsuitable for inclusion in the protocol.
2. Has participated or is participating in any other clinical (investigational) study after completion of CTP2S13031H3 protocol (NCT04072380).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult